CLINICAL TRIAL: NCT03724994
Title: Chemotherapy, Host Response and Molecular Dynamics in Periampullary Cancer
Acronym: CHAMP
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Other Study IDs: CHAMP
Record Dates: First submitted 2018-10-29; First posted 2018-10-30 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Periampullary Adenocarcinoma; Periampullary Cancer; Pancreatic Cancer
Keywords: chemotherapy; adjuvant; palliative; prognostic; predictive; immune response; biomarkers; mutations; cytokines; immune cell signatures
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; folfirinox; Fluorouracil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Plasma samples (for circulating tumor DNA) and serum samples (for cytokines) Tumor cytology and/or tumor biopsy for biomarkers and mutations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study cohort: All patients with periampullary adenocarcinoma or pancreatic cancer receiving palliative or adjuvant chemotherapy (e.g. Gemcitabine, Folfirinox, etc.) in the Department of Oncology, Skåne University hospital, Malmö and Lund
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine — Adjuvant or palliative chemotherapy according to national guidelines
  Other Names: Folfirinox; Gemcitabine - nab-paclitaxel; Fluorouracil; FLOX; 5-FU; 5-Fluorouracil

SUMMARY:
The CHAMP (Chemotherapy, Host response And Molecular dynamics in Periampullary cancer) study is a prospective, single-arm observational study that started Sept 1 2018. Patients diagnosed with pancreatic or other periampullary adenocarcinoma undergoing adjuvant och palliative chemotherapy are invited to participate. The study will examine the tumors' molecular dynamics and how this may change over time and with treatment. Primary endpoint will be overall survival, secondary endpoints will be disease specific survival, time to progression, and quality of life. We estimate that 90 patients will be included in the study per year.

DETAILED DESCRIPTION:
The CHAMP (Chemotherapy, Host response And Molecular dynamics in Periampullary cancer) study is a prospective, single-arm observational study that will start Sept 1 2018. All patients diagnosed with a histologically or cytologically confirmed diagnosis of pancreatic or other periampullary adenocarcinoma undergoing adjuvant or palliative chemotherapy treatment in the Department of Oncology, Skåne University Hospital, Malmö will be invited to participate. The estimated number of recruited patients is 90/year, 75 with pancreatic cancers. Of note tumour origin can seldom be firmly established in non-resectable cases, where only a fine needle aspiration or biopsy specimen is available before initiation of palliative chemotherapy. Main exclusion criteria are: 1. patients having another concomitant life-threatening disease and 2. patients who are unable to receive chemotherapy will be informed about the study by their oncologist and a research nurse and, if they want to participate, will sign an informed consent form.

The treatment regimen will follow national guidelines, and will not be affected by the study. Clinical and pathological data will be compiled at study entry. Radiological and clinical workup will be performed every three months. Primary endpoint will be overall survival, secondary endpoints will be disease specific survival, time to progression, and quality of life (EORTC-QLQ-PAN26). Serial sampling of blood during chemotherapy treatment will be performed by a dedicated research nurse along with the clinical routine sampling. Plasma and serum samples for analysis of ctDNA and cytokines, respectively, will be will be drawn before chemotherapy start (timepoint 0/T0), and prior to each additional course of chemotherapy (monthly e.g. gemcitabine based regimens; T1-5 or biweekly e.g. combination regimen FOLFIRINOX; T1-11), and after the last course of treatment (T6 or T12). Peripheral blood mononuclear cells (PBMC) will be isolated from buffy coat in plasma vials before start of chemotherapy (T0), before the second or third (T2/T3) (monthly or biweekly, respectively) course of chemotherapy, before the fourth or seventh (T4/T7) course of chemotherapy, and after the last course of treatment. A homepage is under construction.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with a histologically or cytologically confirmed diagnosis of pancreatic or other periampullary adenocarcinoma undergoing adjuvant or palliative chemotherapy treatment in the Department of Oncology, Skåne University Hospital, Malmö.

Exclusion Criteria:

1. patients having another concomitant life-threatening disease and
2. patients who are unable to receive chemotherapy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with a histologically or cytologically confirmed diagnosis of pancreatic or other periampullary adenocarcinoma undergoing adjuvant or palliative chemotherapy treatment in the Department of Oncology, Skåne University Hospital, Malmö will be invited to participate.
Sampling Method: Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 years
  months

SECONDARY OUTCOMES:
Time to progression | 5 years
  months
Disease specific survival | 5 years
  months

CONTACTS AND LOCATIONS:
Overall Officials: Karin Jirström, Professor, Study Chair — Lund University; Karin Leandersson, Professor, Study Chair — Lund University; Margareta Heby, MD, Study Chair — Lund University; Sofie Olsson Hau, MD, Study Chair — Lund University
Locations (1):
- Department of Oncology, Skåne University Hospital, Malmo, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Petersson A, Andersson N, Hau SO, Eberhard J, Karlsson J, Chattopadhyay S, Valind A, Elebro J, Nodin B, Leandersson K, Gisselsson D, Jirstrom K. Branching Copy-Number Evolution and Parallel Immune Profiles across the Regional Tumor Space of Resected Pancreatic Cancer. Mol Cancer Res. 2022 May 4;20(5):749-761. doi: 10.1158/1541-7786.MCR-21-0986. PMID 35149544
- [Result] Olsson Hau S, Williamsson C, Andersson B, Eberhard J, Jirstrom K. Sex and gender differences in treatment intention, quality of life and performance status in the first 100 patients with periampullary cancer enrolled in the CHAMP study. BMC Cancer. 2023 Apr 11;23(1):334. doi: 10.1186/s12885-023-10720-w. PMID 37041522
- [Result] Hau SO, Svensson M, Petersson A, Eberhard J, Jirstrom K. Trajectories of immune-related serum proteins and quality of life in patients with pancreatic and other periampullary cancer: the CHAMP study. BMC Cancer. 2023 Nov 7;23(1):1074. doi: 10.1186/s12885-023-11562-2. PMID 37936126
- [Result] Hau SO, Petersson A, Nodin B, Karnevi E, Boman K, Williamsson C, Eberhard J, Leandersson K, Gisselsson D, Heby M, Jirstrom K. Chemotherapy, host response and molecular dynamics in periampullary cancer: the CHAMP study. BMC Cancer. 2020 Apr 15;20(1):308. doi: 10.1186/s12885-020-06807-3. PMID 32293352
- [Derived] Petersson A, Svensson M, Hau SO, Bergstrom R, Lindberg J, Mayrhofer M, Chattopadhyay S, Eberhard J, Heidenblad M, Leandersson K, Gisselsson D, Jirstrom K. Reliable on-treatment prognostication and target identification with a customized assay for circulating tumor DNA in patients with newly diagnosed pancreatic cancer. Sci Rep. 2025 Oct 3;15(1):34481. doi: 10.1038/s41598-025-22369-5. PMID 41044171